CLINICAL TRIAL: NCT03853317
Title: QUILT-3.063: A Phase 2 Study of Combination Therapy With an IL-15 Superagonist (N-803), Off-the-shelf CD16-targeted Natural Killer Cells (haNK), and Avelumab Without Cytotoxic Chemotherapy in Subjects With Merkel Cell Carcinoma (MCC) That Has Progressed on or After Treatment With a Checkpoint Inhibitor.
Brief Title: QUILT-3.063: A Study of N-803, haNK and Avelumab in Patients With Merkel Cell Carcinoma That Has Progressed After Checkpoint Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not meeting recruitment goal
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.063
Record Dates: First submitted 2019-02-14; First posted 2019-02-25 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — avelumab; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with avelumab, haNK™ and N-803 (Experimental): The primary objective is to determine the efficacy of the combination treatment of avelumab, haNK, and N-803 in subjects with MCC that has progressed on or after checkpoint inhibitor therapy by objective response rate (ORR) using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
  Interventions: Biological: Avelumab; Biological: N-803; Biological: haNK™

INTERVENTIONS:
Biological: Avelumab — For the treatment of adults and pediatric patients 12 years and older with Metastatic Merkel Cell Carcinoma (MCC).
  Other Names: (BAVENCIO® injection, for intravenous [IV] use)
Biological: N-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
  Other Names: also known as IL-15N72D:IL-15RαSu/IgG1 Fc complex]), ALT-803
Biological: haNK™ — haNK™ for Infusion is a human, allogeneic, NK cell line that has been engineered to produce endogenous, intracellularly retained IL-2 and to express CD16, the high-affinity (158V) Fc gamma receptor (FcγRIIIa/CD16a).
  Other Names: NK-92 [CD16.158V, ER IL-2], (haNK™ for Infusion)

SUMMARY:
Phase 2, single-arm study to evaluate combination therapy of avelumab, haNK and N-803 in patients with Merkel Cell Carcinoma who have progressed on or after checkpoint inhibitor therapy as assessed by ORR. Patients will receive treatment for a maximum of two years.

DETAILED DESCRIPTION:
This is a phase II, single-arm study of combination therapy of avelumab, haNK, and N-803 in patients with Merkel Cell Carcinoma who have progressed on or after checkpoint inhibitor therapy as assessed by ORR. Patients must have progressed on or within six months of completing treatment with either avelumab or pembrolizumab. Patients will received treatment for a maximum of two years, with avelumab and haNK administered every two weeks, and N-803 administered every three weeks. Radiologic evaluation will occur every eight weeks during the first year of treatment, and every twelve weeks during the second year of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years on day of signing informed consent.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
3. Histologically-confirmed metastatic MCC that has progressed during treatment or within 6 months after completing treatment with single-agent avelumab or pembrolizumab therapy, as per FDA indication.
4. ECOG performance status of 0 to 2.
5. Have at least 1 measurable lesion of ≥ 1.0 cm.
6. Must have a recent FFPE tumor biopsy specimen following the conclusion of the most recent anticancer treatment and be willing to release the specimen for exploratory tumor molecular profiling. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
7. Must be willing to provide blood samples for exploratory analyses.
8. Must be willing to provide a tumor biopsy specimen 8 weeks after the start of treatment for exploratory analyses, if considered safe by the Investigator.
9. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
10. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.

Exclusion Criteria:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
2. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, [subjects with mild rheumatoid arthritis that aren't currently receiving treatment for their disease are eligible for enrollment], Addison's disease, or autoimmune disease associated with lymphoma).
3. History of organ transplant requiring immunosuppression.
4. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
5. Inadequate organ function, evidenced by the following laboratory results:

   1. ANC < 900 cells/mm3.
   2. Platelet count < 75,000 cells/mm3
   3. Total bilirubin greater than twice the ULN (unless the subject has documented Gilbert's syndrome).
   4. AST (SGOT) or ALT (SGPT) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   5. ALP levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
6. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
7. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
8. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
9. Known hypersensitivity to any component of the study medication(s), including anaphylactic reaction to sulfur-containing medications.
10. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
11. Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to the start of treatment on this study, except for testosterone-lowering therapy in men with prostate cancer.
12. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
13. Concurrent participation in any interventional clinical trial.
14. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2022-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Reddy, MD, Study Director — ImmunityBio, Inc.
Locations (5):
- United States (5):
  - University of California San Francisco, San Francisco, California
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Cancer Institute - Baptist Health, Miami, Florida
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Cleveland Clinic Foundation, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Started | 9
Completed | 0
Not Completed | 9
Not completed — Progressive Disease | 5
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — other event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Histologically-confirmed metastatic MCC that has progressed during treatment or within 6 months [Count of Participants; unit: Participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The safety of the combination treatment of avelumab, haNK, and N-803 in subjects with MCC that has progressed on or after checkpoint inhibitor therapy
Time Frame: 30 days after last dose, approximately 1 year 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 9
Participants | 9

2. Primary Outcome: Objective Response Rate
Description: Percent of subjects with confirmed complete Response (CR; disappearance of all target lesions) or partial response (PR; >=30% decrease in the sum of the longest diameter of target lesions) by RECIST v1.1
Time Frame: approximately 1 year 7 months
Measure: Number (95% Confidence Interval); unit: Percent of Subjects
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 9
Percent of Subjects | 0 [0.0 to 33.6]

3. Secondary Outcome: Overall Response Rate by iRECIST (Percent of Subjects With Confirmed Complete or Partial Overall Response)
Description: Percent of subjects with confirmed complete Response (CR; disappearance of all target lesions) or partial response (PR; >=30% decrease in the sum of the longest diameter of target lesions) by iRECIST
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: Percent of Subjects
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 9
Percent of Subjects | 0 [0.00 to 33.6]

4. Secondary Outcome: Progression Free Survival
Description: Defined as the time from the date of first treatment to disease progression or death by any cause, whichever occurs first by RECIST v1.1
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 9
months | 1.9 [1.1 to 1.9]

5. Secondary Outcome: Progression Free Survival
Description: Defined as the time from the date of first treatment to disease progression or death by any cause, whichever occurs first by iRECIST
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 9
Months | 1.9 [1.1 to NA] — Due to the small number of subjects an upper bound on the confidence interval was not able to be calculated

6. Secondary Outcome: Overall Survival
Description: Overall Survival defined as the time from the date of first treatment to death by any cause
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 9
months | 5.6 [1.1 to NA] — Due to the small number of subjects an upper bound on the confidence interval was not able to be calculated

7. Secondary Outcome: Disease-Specific Survival
Description: Disease-Specific Survival defined as the time from the date of first treatment to death resulting from MCC
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 9
months | NA [1.9 to NA] — Due to the small number of subjects the median disease-specific survival and the upper bound on the confidence interval were not able to be calculated

8. Secondary Outcome: Disease Control Rate
Description: Percent of subjects with stable disease for >= 8 weeks, or confirmed complete Response (CR; disappearance of all target lesions) or partial response (PR; >=30% decrease in the sum of the longest diameter of target lesions) by RECIST v1.1
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: Percent of Subjects
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 9
Percent of Subjects | 0.00 [0.00 to 33.6]

9. Secondary Outcome: Disease Control Rate
Description: Percent of subjects with stable disease for >= 8 weeks, or confirmed complete Response (CR; disappearance of all target lesions) or partial response (PR; >=30% decrease in the sum of the longest diameter of target lesions) by iRECIST
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: Percent of Subjects
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 9
Percent of Subjects | 0 [0.00 to 33.6]

10. Secondary Outcome: FACT-M Total Score
Description: Quality of Life Measures as measured by the Functional Assessment of Cancer Therapy-Melanoma (FACT-M) instrument's FACT-M Total Score. The FACT-M total score is a sum of the questions from its six subscales (a sum of 51 questions in total): Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Additional Concerns, and At the Site of Melanoma. All subscale questions use a 5-point Likert-type response score ranging from 0 = 'not at all' to 4 = 'very much'. The FACT-M Total score, therefore, ranges from 0 to 204. Negatively worded items are reverse scored prior to summing so that higher subscale and total scores indicate a better quality of life
Time Frame: Baseline, Week 13, and End of Treatment visit, up to 2 years
Population: At week 13 only 2 subjects had quality of life measurements. At end of treatment only 5 subjects had quality of life measurements.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 9
Scores on a scale
  Baseline | 143.8 (26.55)
  Week 13: number analyzed (Participants) | 2
  Week 13 | 144.5 (13.44)
  End of Treatment: number analyzed (Participants) | 5
  End of Treatment | 126.6 (31.55)

11. Secondary Outcome: Duration of Response by RECIST Version 1.1 and iRECIST
Description: Duration of Response is defined as the time from the date of first response (Investigator-assessed PR or CR) to the date of disease progression or death (any cause) whichever occurs first. Per RECIST and iRECIST: a complete response is the disappearance of all target lesions; a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From time of CR or PR up to 2 years
Population: No subject had a complete or partial response
Arm/Group | Treatment With Avelumab, haNK™ and N-803
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days after last dose, up to 2 years or until resolution or stabilization for nonserious grade 3 or 4 AEs and SAEs, whichever is longer.
Arm/Group | Treatment With Avelumab, haNK™ and N-803
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Avelumab, haNK™ and N-803 (N=9)
Anaemia (Blood and lymphatic system disorders) | 2
Oedema peripheral (General disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Haematuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Avelumab, haNK™ and N-803 (N=9)
Chills (General disorders) | 5
pyrexia (General disorders) | 4
fatigue (General disorders) | 2
Injection site erythrma (General disorders) | 2
Injection site pruritus (General disorders) | 2
Injection site reaction (General disorders) | 2
asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Eosinophilia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 2
Proteinuria (Renal and urinary disorders) | 2
Chromaturia (Renal and urinary disorders) | 1
Glycosuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3
Wound complication (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Candida infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT03853317/Prot_SAP_000.pdf